CLINICAL TRIAL: NCT02252575
Title: Assessment of Electromagnetic Interference Between E-transportation and Cardiac Implantable Electronic Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-014
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Electromagnetic Interference
MeSH Terms: interventions — Magnetic Field Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electromagnetic field (Experimental): Exposure to the elctromagnetic field of an electric motor
  Interventions: Device: Electromagnetic field

INTERVENTIONS:
Device: Electromagnetic field — Exposure to the electromagnetic fields of electric motors

SUMMARY:
E-Transportation is increasing all over the world. It is not known if the used engines interfere with cardiac implantable electronic devices. The study evaluates such potential interferences in vivo.

DETAILED DESCRIPTION:
E-Transportation is increasing all over the world. It is not known if the used engines interfere with cardiac implantable electronic devices. The study evaluates different types of electric motors with regard to electromagnetic interference with implanted pacemakers or cardioverter-defibrillators.

ELIGIBILITY:
Inclusion Criteria:

* implanted cardiac implantable electronic device with regular function

Exclusion Criteria:

* implanted cardiac implantable electronic device with irregular function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of electromagnetic interference | acute setting
  Occurrence of electromgantic interference during an exposure time of approximately 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kolb, MD, Study Chair — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany